CLINICAL TRIAL: NCT06673238
Title: A First-In-Human Study to Evaluate the Pharmacokinetics, Safety, and Tolerability of ABBV-722 Following Single and Multiple Ascending Doses in Healthy Adult Subjects and Single Doses in Healthy Adult Asian Subjects
Brief Title: A Study to Assess How the Drug Moves Through the Body, Adverse Events, and Tolerability of Oral ABBV-722 Capsules of Single and Multiple Ascending Doses in Adult Participants and Single Doses in Adult Asian Participants
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: M25-150
Record Dates: First submitted 2024-10-29; First posted 2024-11-04 (Actual); Last update posted 2025-07-20 (Actual); Status verified 2025-07

CONDITIONS: Healthy Volunteer
Keywords: Healthy Volunteer; ABBV-722

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (12):
- Part 1: Group 1 (Experimental): Participants will receive a single dose of either ABBV-722 Dose A or placebo.
  Interventions: Drug: ABBV-722; Drug: Placebo
- Part 1: Group 2 (Experimental): Participants will receive a single dose of either ABBV-722 Dose B or placebo.
  Interventions: Drug: ABBV-722; Drug: Placebo
- Part 1: Group 3 (Experimental): Participants will receive a single dose of either ABBV-722 Dose C or placebo.
  Interventions: Drug: ABBV-722; Drug: Placebo
- Part 1: Group 4 (Experimental): Participants will receive a single dose of either ABBV-722 Dose TBD or placebo.
  Interventions: Drug: ABBV-722; Drug: Placebo
- Part 1: Group 5 (Experimental): Participants will receive a single dose of either ABBV-722 Dose TBD or placebo.
  Interventions: Drug: ABBV-722; Drug: Placebo
- Part 2: Group 6 (Experimental): Participants who are Han Chinese will receive a single dose of ABBV-722 Dose D.
  Interventions: Drug: ABBV-722
- Part 2: Group 7 (Experimental): Participants who are Japanese will receive a single dose of ABBV-722 Dose D.
  Interventions: Drug: ABBV-722
- Part 3: Group 8 (Experimental): Participants will receive either ABBV-722 Dose E or placebo for 14 days.
  Interventions: Drug: ABBV-722; Drug: Placebo
- Part 3: Group 9 (Experimental): Participants will receive either ABBV-722 Dose F or placebo for 14 days.
  Interventions: Drug: ABBV-722; Drug: Placebo
- Part 3: Group 10 (Experimental): Participants will receive either ABBV-722 Dose A or placebo for 14 days.
  Interventions: Drug: ABBV-722; Drug: Placebo
- Part 3: Group 11 (Experimental): Participants will receive either ABBV-722 Dose G or placebo for 14 days.
  Interventions: Drug: ABBV-722; Drug: Placebo
- Part 3: Group 12 (Experimental): Participants will receive either ABBV-722 Dose TBD or placebo for 14 days.
  Interventions: Drug: ABBV-722; Drug: Placebo

INTERVENTIONS:
Drug: ABBV-722 — Oral Capsule
Drug: Placebo — Oral Capsule
  Arms: Part 1: Group 1; Part 1: Group 2; Part 1: Group 3; Part 1: Group 4; Part 1: Group 5; Part 3: Group 10; Part 3: Group 11; Part 3: Group 12; Part 3: Group 8; Part 3: Group 9

SUMMARY:
This is a Phase 1, first-in-human study to investigate safety, tolerability, and pharmacokinetics of ABBV-722 after oral dosing in healthy adult participants.

ELIGIBILITY:
Inclusion Criteria:

* Laboratory values meet the criteria specified in the protocol.
* A condition of general good health, based upon the results of a medical history, physical examination, vital signs, laboratory profile, and a 12-lead electrocardiogram (ECG).
* Part 2 only: Healthy Han Chinese and Japanese individuals between 18 and 65 years of age, inclusive at the time of Screening.

  * Participant must be first- or second-generation Han Chinese of full Chinese parentage (both parents of Han Chinese descent), residing outside of China. Participants must be in general good health and maintain a typical Chinese lifestyle, including consuming a typical Chinese diet.
  * First-generation participants will have been born in China to two parents and four grandparents, who were also born in China, and are of full Chinese descent.
  * Second-generation participants born outside of China must have two parents and four grandparents born in China and are of full Chinese descent. OR
  * Participant must be first- or second-generation Japanese of full Japanese parentage (both parents of Japanese descent), residing outside of Japan. Participants must be in general good health and maintain a typical Japanese lifestyle, including consuming a typical Japanese diet.
  * First-generation participants will have been born in Japan to two parents and four grandparents, who were also born in Japan, and are of full Japanese descent.
  * Second-generation participants born outside of Japan must have two parents and four grandparents born in Japan and are of full Japanese descent.

Exclusion Criteria:

* History of any clinically significant illness/infection/major febrile illness, hospitalization, or any surgical procedure within 30 days prior to the first dose of study drug.
* Consumption of alcohol, grapefruit products, Seville oranges, starfruit products or quinine/tonic water within the 72-hour period prior to study drug administration.
* Use of tobacco or nicotine-containing products within 180 days prior to the first dose of study drug.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 96 (Estimated)
Dates: Start 2024-10-29 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with Adverse Events Reported During Safety Evaluations | Up to Day 44
  Safety evaluations will include AE monitoring, vital sign measurements (including orthostatic blood pressure and pulse rate), ECG variables, and clinical laboratory testing (hematology, chemistry, and urinalysis) as a measure of safety and tolerability for the entire study duration. Clinically significant abnormal changes in physical examination findings will be reported as AEs.
Maximum Plasma Concentration (Cmax) of ABBV-722 | Up to Day 21
  Cmax of ABBV-722.
Time to Cmax (Tmax) of ABBV-722 | Up to Day 21
  Tmax of ABBV-722.
For Parts 1 and 2: Area Under the Concentration-Time Curve (AUC) from Time 0 to Time t (AUCt) of ABBV-722 | Up to Day 8
  AUCt of ABBV-722.
For Parts 1 and 2: Area Under the Concentration-Time Curve (AUC) from Time 0 to Infinity (AUCinf) of ABBV-722 | Up to Day 8
  AUCinf of ABBV-722
For Part 3: Observed Plasma Concentration at the End of the Dosing Interval (Ctrough) of ABBV-722 | Up to Day 21
  Ctrough of ABBV-722.
For Part 3: AUC from Time 0 to the End of Dosing Interval (AUCtau) Following the First and Last Doses of ABBV-722 | Up to Day 21
  AUC from AUCtau following the first and last doses of ABBV-722.
Terminal Phase Elimination Rate Constant (Beta) of ABBV-722 | Up to Day 21
  Beta of ABBV-722.
Terminal Phase Elimination Half-Life (t1/2) of ABBV-722 | Up to Day 21
  t1/2 of ABBV-722.
Dose Normalized Cmax | Up to Day 21
  Dose normalized Cmax.
Dose Normalized AUCs | Up to Day 21
  Dose normalized AUCs.

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (1):
- Acpru /Id# 270279, Grayslake, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Related Info — https://www.abbvieclinicaltrials.com/study/?id=M25-150